CLINICAL TRIAL: NCT03884049
Title: Novel Transcatheter Arterial Embolization for Treatment of Knee Osteoarthritis: a Randomized Sham-controlled Clinical Trial
Brief Title: Neovascularization Embolisation for Knee Osteoarthritis.(NEO)
Acronym: NEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: William Cook Europe (Industry); Stichting Coolsingel (Unknown)
Responsible Party: Principal Investigator, Dr. Edwin Oei, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METC 2018-081; 2018-081 (Registry Identifier: METC ErasmusMC)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee
Keywords: ranscatheter; embolization; osteoarthritis; arterial
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Embolization, Therapeutic

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized placebo-controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embolization group (Experimental): Group undergoes transcatheter arterial embolization of neovessels around the knee.
  Interventions: Procedure: Embolization
- Sham Embolization Group (Sham Comparator): Group undergoes sham embolization
  Interventions: Procedure: Sham embolization

INTERVENTIONS:
Procedure: Embolization — transcatheter arterial embolization of neovessels around the knee
  Arms: Embolization group
Procedure: Sham embolization — Sham transcatheter arterial embolization of neovessels in the knee
  Arms: Sham Embolization Group

SUMMARY:
In this double blind randomized sham controlled study the investigators want to establish the efficacy of transcatheter arterial embolization of neovessels for patients with symptomatic mild to moderate knee osteoarthritis after 4 months compared to a sham-embolization.

DETAILED DESCRIPTION:
Rationale:

Transcatheter arterial embolization has recently been proposed as an efficacious therapy for therapy-resistant osteoarthritis of the knee, providing substantial pain reduction at short-term as well as long-term follow-up up till 4 years.

A potential working mechanism of treatment effect is that the normalization of the amount of blood vessels and blood flow achieved by embolization reduces inflammation, resulting in pain reduction

Objective:

The main objective is to assess whether transcatheter arterial embolization of neovessels in patients with symptomatic knee OA results in significant pain reduction after 4 months compared to sham treatment.

The investigators hypothesize that novel transcatheter arterial embolization of neovessels is a feasible, effective, and safe treatment for patients with symptomatic radiographic knee OA, resulting in significant improvement of pain symptoms in a period of 4 months follow-up compared to sham embolization.

Secondary objectives are

1. to assess whether reduction of neovessels is related to pain relief,
2. to explore whether decrease of inflammation is a mediating factor between neovessel reduction and pain relief,
3. to assess whether transcatheter arterial embolization reduction of neovessels decreases peripheral and central pain sensitization and
4. to assess whether transcatheter arterial embolization improve the outcome at 1, 4, 8 and 12 months compared to placebo of the: ICOAP, painDETECT, EQ-5D-5L questionnaires and NRS for pain.

ELIGIBILITY:
Inclusion Criteria:

* Age.≥18 years
* Knee pain for a duration of ≥ 6 months
* Knee pain (numeric rating scale ≥4 - ≤8) on at least half of the days in the preceding month at time of inclusion.
* There is insufficient response of conservative treatment for at least 6 months
* Radiographic knee osteoarthritis (radiographic Kellgren and Lawrence grade 1-3)

Exlusion criteria:

* Contra-indications for MRI (e.g. metallic foreign bodies, etc.)
* Contra-indications for angiography
* Renal insufficiency, checked with blood sample test (GFR < 30 ml/min/1, 73 m2);
* Known allergy to contrast agents;
* Patient has known allergies to barium sulfate, 3-aminopropyltrialkoxysilane, polyphosphazene
* Women who are pregnant or lactating
* Intermittent claudication of affected limb
* Intra articular injections in the ipsilateral knee less than 6 months ago
* On the waiting list for joint replacement surgery
* Amitriptyline usage.
* Patient has known allergies to barium sulfate, 3-aminopropyltrialkoxysilane, polyphosphazene.
* Insufficient command of the Dutch or English language.
* Legally incompetent adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
KOOS pain sub score | 4 months
  KOOS pain sub score after 4 months

SECONDARY OUTCOMES:
Total KOOS | 1,4,8,12 month(s)
  Total KOOS result
painDETECT questionnaire | 1,4,8,12 month(s)
  painDETECT questionnaire results
ICOAP questionnaire | 1,4,8,12 month(s)
  ICOAP questionnaire results
Pain Score 0-10 Numerical Rating Scale (NRS) | 1,4,8,12 month(s)
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
EQ-5D-5L questionnaire | 1,4,8,12 month(s)
  EQ-5D-5L questionnaire results
Pressure pain threshold testing | 1,4,8,12 month(s)
  Pressure pain threshold testing results
Knee MRI | 1 and 4 month(s)
  Knee MRI scan results

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Edwin, MD, PhD, Principal Investigator — Erasmus Medical Center; Adriaan Moelker, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We are willing the share all our available unidentified data on reasonable request
Supporting Information: Study Protocol
Time Frame: is available upon request as of now and will be available for the next 15 years.
Access Criteria: * after written request to PI
  * after signing Data Transfer Agreement
  * No commercial use for data allowed by requesting party.

REFERENCES:
- [Derived] van Zadelhoff TA, Bos PK, Moelker A, Bierma-Zeinstra SMA, van der Heijden RA, Oei EHG. Genicular artery embolisation versus sham embolisation for symptomatic osteoarthritis of the knee: a randomised controlled trial. BMJ Open. 2024 Oct 1;14(10):e087047. doi: 10.1136/bmjopen-2024-087047. PMID 39353688
- [Derived] van Zadelhoff TA, Moelker A, Bierma-Zeinstra SMA, Bos PK, Krestin GP, Oei EHG. Genicular artery embolization as a novel treatment for mild to moderate knee osteoarthritis: protocol design of a randomized sham-controlled clinical trial. Trials. 2022 Jan 8;23(1):24. doi: 10.1186/s13063-021-05942-x. PMID 34998425